CLINICAL TRIAL: NCT04391413
Title: Does Optical Coherence Tomography Optimise Results of Stenting of the Left Main Stem
Brief Title: Does OCT Optimise Results of Stenting on the Left Main Stem
Acronym: DOCTORS-LM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A00532-37
Record Dates: First submitted 2020-04-02; First posted 2020-05-18 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Myocardial Infarction; Myocardial Ischemia; Non ST Segment Elevation Myocardial Infarction
Keywords: left main stem; angioplasty; optical coherence tomography; myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OCT group (Experimental): OCT will be performed after initial coronary angiography and at the end of the procedure. Several OCT runs can be performed. The operator may change procedural strategy, and use additional interventions. The operator must evaluate the following parameters, based on OCT data:
  Before angioplasty: reference diameter and reference area of distal main vessel; lesion length; presence and extent of thrombus or calcification.
  Stent implantation: Stent should be sized according to distal reference diameter, and should allow for expansion to the reference diameter of the proximal main vessel.
  After stent implantation: minimal and reference lumen diameter, minimal and reference lumen area, minimal stent area, presence of thrombus, presence of edge dissection, tissue protrusion, optimal lesion coverage, malapposition, suboptimal stent deployment.
  Interventions: Device: Use of OCT to guide the angioplasty procedure
- Control group (No Intervention): Angioplasty will be guided by traditional fluoroscopy alone, performed before and after stent implantation. The recommendation for angioplasty of left main stenosis is to use main vessel (MV) stenting with a proximal optimisation technique (POT) and provisional side branch (SB) stenting as a preferred approach. Predilatation of the side branch (SB) may be considered, but is recommended in the following circumstances: extensive ostial SB involvement, heavy calcification, etc. even with a provisional SB stenting approach.

INTERVENTIONS:
Device: Use of OCT to guide the angioplasty procedure — OCT will be performed and OCT data used to choose and/or modify procedural strategy. The OCT system used will be the Ilumien Optis system, and Dragonfly Optis probe.
  Arms: OCT group

SUMMARY:
The DOCTORS-LM study will investigate the impact of using optical coherence tomography (OCT) to guide the procedure in angioplasty of lesions of the left main stem responsible for myocardial ischemia.

DETAILED DESCRIPTION:
Angiographic evaluation of lesions of the left main stem presents particular challenges and high procedural complexity. The clinical sequelae of a suboptimal result in this context may be severe, and thus, it is recommended that patients with left-main lesions be considered for imaging-guided interventions by means of optimal coherence tomography (OCT) in non-ostial left main lesions. The investigators have previously demonstrated in a randomized trial of patients undergoing PCI for a lesion responsible for non ST elevation acute coronary syndromes that OCT provides useful clinical information beyond that obtained by angiography alone, and OCT-guidance for angioplasty in these patients yielded a significantly higher proportion of patients with an optimal functional result after stenting. In this context, the aim of the present study is to evaluate whether OCT-guided left-main angioplasty is superior to left main angioplasty guided by fluoroscopy alone, as assessed by fractional flow reserve (FFR) measured after stent implantation. Eligible patients must be aged 18 years and over, admitted for acute coronary syndrome (ACS) or stable coronary artery disease (CAD); AND present an angiographically significant non-ostial lesion of the left main stem requiring angioplasty with drug eluting stent implantation.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 years or over presenting with:

* NSTEMI or unstable angina or stable angina or documented silent ischemia AND
* De novo angiographic lesion (% diameter stenosis >=50%) or functionally significant (FFR<=0.80) lesion of the left main stem (median or distal) with or without lesions of the ostia of the LAD and/or circumflex arteries (= Medina classification 1-0-0, 1-0-1, 1-1-0, 1-1-1) or ostial lesion of the LAD and/or circumflex artery requiring angioplasty with stent implantation that will cover the distal left main stem (=Medina classification 0-0-1, 0-1-0 ou 0-1-1) AND
* SYNTAX score ≤ 22 (or >22 and ≤32 and validated by the Heart Team)
* Lesion with reference angiographic diameter <=5.5mm
* Signature of written informed consent form.

Exclusion Criteria:

Patients with:

* ST segment elevation myocardial infarction
* Ostial lesion of the left main stem
* Technically impossible to perform OCT
* Creatinine clearance ≤ 30 ml/min/1.73m²
* Left ventricular ejection fraction <30%
* Hypotension or cardiogenic shock
* Unstable ventricular arrhythmia
* Contraindication to dual antiplatelet therapy for at least 6 (or 12) months (duration depending on the initial clinical presentation). Shorter dual antiplatelet therapy is possible in patients with long-term anticoagulation.
* Hypersensitivity or contraindication to any of the antithrombotic therapies used during or after the procedure
* Life expectancy <1 year
* Persons under judicial protection
* Subjects with no social security coverage
* Anticipated non-compliance with the study procedures
* Pregnant or lactating women
* Subjects within the exclusion period of another clinical trial
* Failure to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2023-07-16 (Estimated)

PRIMARY OUTCOMES:
Functional outcome of the procedure (absolute value) | At the end of the procedure, once the operator judges the result to be satisfactory.
  Functional outcome as assessed by the Fractional flow reserve (FFR) at the end of the procedure (average of at least 3 consecutive measures)

SECONDARY OUTCOMES:
Functional outcome of the procedure (dichotomized) | At the end of the procedure, once the operator judges the result to be satisfactory.
  Percentage of patients with a final fractional flow reserve (FFR) value >=0.90
Relative change in final FFR value | At the end of the angioplasty procedure
  Relative change in final FFR value as compared to initial FFR value at the start of the procedure in each patient
Percentage of patients in whom OCT after stent implantation reveals a suboptimal result | Immediately after stent implantation
  Percentage of patients in whom OCT after stenting reveals a sub-optimal result, defined as the presence of any one or more of the following criteria:
  * Stent under expansion
  * Stent malapposition
  * Lesion incompletely covered by the stent
  * Residual stenosis upstream or downstream of the stent
  * Edge dissection
  * Thrombus
  * Tissue protrusion through the stent struts
Percentage of patients in whom a change in procedural strategy is decided based on OCT data | Immediately after stent implantation
  Percentage of patients in whom a change in procedural strategy is decided based on OCT data, with use of any one or more of the following:
  * GPIIb/IIIa inhibitors
  * Thrombo aspiration
  * Rotational atherectomy
  * Additional stent implantation
  * Additional balloon inflations
  * Re-opening of strent struts in secondary branch
Safety of OCT in angioplasty of the left main stem | At the end of the angioplasty procedure
  Safety of OCT in angioplasty of the left main stem, as assessed by duration of procedure (minutes)
Safety of OCT in angioplasty of the left main stem | At the end of the angioplasty procedure
  Safety of OCT in angioplasty of the left main stem, as assessed by - fluoroscopy time (minutes)
Safety of OCT in angioplasty of the left main stem | At the end of the angioplasty procedure
  Safety of OCT in angioplasty of the left main stem, as assessed by Radiation dose received (MSv)
Safety of OCT in angioplasty of the left main stem | At the end of the angioplasty procedure
  Safety of OCT in angioplasty of the left main stem, as assessed by Quantity of contrast medium used (mL)
Safety of OCT in angioplasty of the left main stem | At the end of the angioplasty procedure
  Safety of OCT in angioplasty of the left main stem, as assessed by change in creatinine clearance over the first 24 hours (Creatinine clearance in ml/min)
Safety of OCT in angioplasty of the left main stem | At the end of the angioplasty procedure
  Safety of OCT in angioplasty of the left main stem, as assessed by procedural complications
OCT data that predict final FFR value >=0.90 | At the end of the angioplasty procedure
  Thresholds for minimal lumen diameter and minimal stent area on OCT that best predict a final FFR value >=0.90

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Meneveau, MD, PhD, Principal Investigator — Cardiology Department, CHU Besancon
Locations (12):
- France (12):
  - CHU Besancon, Besançon, Please Select
  - CHRU Lille, Lille, Please Select
  - Hôpital Privé Saint Martin, Caen
  - Centre Hospitalier de Chartres - Hôpital Louis Pasteur, Chartres
  - CHRU Clermont Ferrand, Clermont-Ferrand
  - Institut Cardiovasculaire Paris Sud, Massy
  - CHU Nîmes - Hôpital Carémeau, Nîmes
  - Institut Mutualiste Montsouris, Paris
  - CHU Poitiers, Poitiers
  - Clinique Saint Hilaire, Rouen
  - Institut Arnault Tzanck, Saint-Laurent-du-Var
  - Hôpital Nord Franche-Comté, Trévenans

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meneveau N, Souteyrand G, Motreff P, Caussin C, Amabile N, Ohlmann P, Morel O, Lefrancois Y, Descotes-Genon V, Silvain J, Braik N, Chopard R, Chatot M, Ecarnot F, Tauzin H, Van Belle E, Belle L, Schiele F. Optical Coherence Tomography to Optimize Results of Percutaneous Coronary Intervention in Patients with Non-ST-Elevation Acute Coronary Syndrome: Results of the Multicenter, Randomized DOCTORS Study (Does Optical Coherence Tomography Optimize Results of Stenting). Circulation. 2016 Sep 27;134(13):906-17. doi: 10.1161/CIRCULATIONAHA.116.024393. Epub 2016 Aug 29. PMID 27573032